CLINICAL TRIAL: NCT03281798
Title: Fetal Cystoscopy for Severe Lower Urinary Tract Obstruction (LUTO): A Prospective Trial
Brief Title: Fetal Cystoscopy for Severe Lower Urinary Tract Obstruction
Acronym: CYSTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Ruano (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Ruano, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220117-1; 16-008556 (Other: Mayo Clinic); NCT05368727 (obsolete NCT alias)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Lower Urinary Tract Obstructive Syndrome; Lower Urinary Tract Obstruction, Congenital; Bladder Outlet Obstruction; Bladder Outflow Obstruction
MeSH Terms: conditions — Urinary Bladder Neck Obstruction | interventions — Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fetal Cystoscopy Group (Experimental): Participants in this group will receive the fetal cystoscopy procedure around 16 weeks 0 days to 25 weeks and 6 days of gestation.
  Interventions: Device: Fetoscopes; Procedure: Fetal Cystoscopy

INTERVENTIONS:
Device: Fetoscopes — Fetoscopes are telescopes developed for procedures involving fetal interventions and is inserted through the maternal abdomen.
Procedure: Fetal Cystoscopy — A fetoscope will be inserted into the fetal bladder via the maternal abdomen and advanced into the fetal bladder outlet. Identified obstruction will be opened using laser.

SUMMARY:
The purpose of the study is to study the outcomes of maternal and fetal patients who are undergoing fetal intervention for severe isolated lower urinary tract obstruction (LUTO).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women
2. Singleton pregnancy
3. Maternal age ≥ 18 years
4. Male fetus with LUTO, dilated bladder, "keyhole sign" and bilateral hydronephrosis
5. Oligohydramnios or Anhydramnios
6. Favorable urine analysis defined as urinary sodium is < 100 milliequivalents per liter (mEq/L), chloride < 90 mEq/L, and osmolality < 200 milliosmoles per kilogram (mOsm/kg) after 20 weeks and in the absence of previous in utero intervention for the disease (vesicoamniotic shunt placement or fetal cystoscopy).
7. Absence of chromosomal abnormalities and associated anomalies
8. Gestational age at the time of the procedure will be between 16 0/7 weeks and 25 6/7 weeks
9. Normal karyotype by invasive testing (amniocentesis or Chorionic Villus Sampling (CVS)). Patients declining invasive testing will be excluded.
10. Family have considered and declined the option of termination of the pregnancy at less than 24 weeks.
11. Family meets psychosocial criteria, including sufficient social support and ability to understand requirements of the study.
12. Parents or guardian are willing to provide signed informed consent.

Exclusion Criteria:

1. Fetal anomaly unrelated to LUTO
2. Congenital cardiac anomaly
3. Female fetus
4. Increased risk for preterm labor including short cervical length (<1.5 cm), history of incompetent cervix with or without cerclage, and previous preterm birth
5. Placental abnormalities (previa, abruption, accreta) known at time of enrollment
6. Contraindications to surgery including previous hysterotomy in active uterine segment
7. Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, uterine anomalies incompatible with fetoscopy
8. Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
9. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
10. Maternal medical condition that is a contraindication to surgery or anesthesia
11. Patient does not have health insurance to cover routine clinical care including prenatal care, prenatal ultrasound, amniocentesis, tocolysis, admission, delivery, and fetal vesico-amniotic shunting. The exception will be fetal cystoscopy which is considered an experimental procedure.
12. Inability to comply with travel and follow-up requirements of the trial
13. Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy
14. Patients declining invasive testing
15. Family does not meet psychosocial criteria including insufficient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants where the procedure was technically performed | Day 1 (Post fetal cystoscopy procedure)
  Number of participants where the fetal cystoscopy procedure was successfully technically performed.
Number of participants where the etiology of LUTO was correctly diagnosed | Up to 1 month post delivery
  Number of participants where the etiology of LUTO was correctly diagnosed during fetal cystoscopy as compared to post natal cystoscopy
Number of participants where the posterior urethral valve were successfully released | Day 1 (Post fetal cystoscopy procedure)
  Number of participants where the posterior urethral valve were successfully released
Number of participants whose fetal cystoscopy resulted in the prevention of post-natal severe pulmonary hypoplasia | Up to 1 month post delivery
  As per treating physician evaluation of clinical assessments post-natal.
Number of participants whose fetal cystoscopy resulted in the prevention of post-natal severe renal impairment | Up to 24 months post delivery
  As per treating physician evaluation of clinical assessments post-natal.
Number of participants whose fetal cystoscopy resulted in maternal complications | Day 1 post delivery
  Maternal and obstetrical complications such as preterm premature rupture of the membranes (PPROM), prematurity (birth <37 weeks), extremely preterm birth (<32 weeks), and urological fistulae and fetal demise.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD, PhD., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No